CLINICAL TRIAL: NCT05984316
Title: The Effect of Exercises Applied With Dual-Duty Approach on Physical and Cognitive Status in Cases With Juvenile-Onset Systemic Lupus Erythematosus
Brief Title: Systemic Lupus Erythematosus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Eylül Pınar KISA, PHD, Biruni University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLE
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: System; Lupus Erythematosus; Cognition Disorder; Autoimmune
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Cognition Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise group (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Dual task exercises are defined as the appropriate direction of attention during two activities performed at the same time. Dual task performance is required during many activities in daily life. Multitasking is complicated to understand because it is divided into social, physical, and psychological branches.
  The simultaneous occurrence of movement and cognitive processes is seen as a part of social participation. Considering that one task affects the other, dual task is defined as the simultaneous performance of two tasks that can be performed independently, can be evaluated separately, and have different purposes.
  Each task must be incompatible and measurable, achievable alone or in different combinations. The increased need for information processing alone does not constitute dual-tasking.

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic autoimmune and inflammatory disease. The pathogenesis of SLE results from interactions between genes, hormones, and the environment; however, the exact etiology is unknown. SLE can affect many organs and systems, including the musculoskeletal, hematological, renal, neuropsychiatric, cardiovascular and pulmonary systems, and skin. Non-specific general complaints such as malaise, fatigue, arthralgia, anxiety, depression, fever, and weight loss are evident at the onset of the disease and during the activation periods. Patients experience hopelessness due to the complexity of the symptoms and the chronic and progressive nature of the disease, and they experience deterioration in their quality of life due to the interaction of anxiety and depression findings with other symptoms. SLE is a difficult disease to manage because of the different organ and system involvement processes.

In addition, these symptoms of the disease and the nature of chronic pain, including central sensitization, cause it to accompany a process that is affected by the mood of the person. Some patients present to a rheumatologist with mild symptoms, while others may present with severe, life-threatening symptoms. The onset of the disease before the age of 18 is defined as childhood onset (juvenile). Childhood-onset SLE accounts for approximately 1/5 of SLE patients. It is known that the main mechanism in the formation of the disease is the production of more than one autoantibody.

Although childhood SLE (jSLE) appears to be basically the same disease with similar etiology, pathogenesis, and laboratory findings as in adults, there are differences in the frequency and severity of clinical manifestations. In this respect, the clearest finding is that children with SLE have greater disease severity and earlier disease-related organ damage than adults with SLE. Studies on the disease show that patients with jSLE have not only physical but also cognitive effects.

The aim of our study is to examine the effects of exercises applied with a dual-task approach on patients' physical and cognitive status in jSLE cases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 6-16 years diagnosed with jSLE by a pediatric rheumatologist
2. Those who have had the disease for at least one year
3. Those whose medical treatments are in a stable period
4. Patients willing to be rehabilitated and able to adapt to the study

Exclusion Criteria:

1. Cases older than 16 years old diagnosed with jSLE
2. Patients with initiation of multi-organ failure
3. Those whose medical treatments are in flux
4. Wanting to leave the study
5. Not participating in assessments
6. Not attending treatment programs regularly
7. Not being able to adapt to treatment programs at the cognitive level

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2023-12-02 (Estimated); Study Completion 2023-12-05 (Estimated)

PRIMARY OUTCOMES:
Cognitive eveluation | 0-16. week
  Children's cognitive level will be evaluated with the Montreal Cognitive Assessment (MoCA), a rapid screening test for mild cognitive impairment. MoCA assesses different cognitive functions. These; attention and concentration, executive functions, memory, language, visual construction skills, abstract thinking, calculation and orientation. MoCA takes about 10 minutes to apply. The highest total score that can be obtained from the test is 30. Accordingly, a score of 21 points or more is considered normal.

SECONDARY OUTCOMES:
Pain assessment | 0-16. week
  Part One: There are 15 descriptive word groups in this part. Of these, 11 evaluate the sensory dimension of the pain, and 4 evaluate the perceptual dimension. These descriptors are rated on an intensity scale from 0 to 3 (0= none, 1= Mild, 2=Moderate, 3= Excess). In the first part of the scale, a total of 3 pain scores are obtained: sensory pain score, perceptual pain score and total pain score.
  Part Two: In the second part of the form, there are five word groups ranging from "mild pain" to "unbearable pain" to determine the severity of the patient's pain.
  In Part Three: In the third part, the patient's current pain intensity is evaluated using a visual comparison scale.
Disease activity | 0-16. week
  Disease activity of children will be evaluated with the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI). Originally defined in 1992, SLEDAI is a global index of 24 clinical and laboratory variables with distinct differences reflecting disease activity over the past 10 days. Neurological, locomotor, renal, The activity is evaluated in nine systems: mucocutaneous, general, cardiac, respiratory, vascular, and haematological. The maximum score is 105.
Activity Assessment | 0-16. week
  It consists of two different parts, the disability index and the discomfort index. Disability index dressing and It consists of 8 parameters including self-care, standing up, eating, walking, hygiene, reaching, holding and activities. A non-applicable answer is available for each question to eliminate bias due to age and growth limitations. The representation score is calculated according to the highest scores answered in that area. Discomfort is assessed by measuring pain with a 15 cm visual analog scale. Parents of the patients told their children's last week A VAS score is made about how much pain they have inside and they are asked to give a score between 0 and 100. Likewise, they are asked to score between 0 and 100 on how much they have been affected by the disease since the onset of the disease. The CHAQ score is calculated by adding the disability and discomfort scores and then dividing by 2. The higher the score, the worse the child's condition.
Physical activity assessment | 0-16 weeks
  The physical activity levels of the subjects participating in the study It will be followed by a smart wristband with a physical activity monitor at the beginning and during the training sessions.

CONTACTS AND LOCATIONS:
Overall Officials: eylul Pinar kısa, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kisa EP, Sahin S, Leblebici G, Tonyali IY, Balci G, Dilek S, Aslan E, Tarakci E, Kasapcopur O. Effects of dual-task exercises on cognitive status, disease activity and quality of life in childhood-onset systemic lupus erythematosus. Lupus Sci Med. 2025 Jun 19;12(1):e001453. doi: 10.1136/lupus-2024-001453. PMID 40541266